CLINICAL TRIAL: NCT03535597
Title: A Randomized Comparison of the QuikClot® Radial® Pad Versus the Standard of Care TR Band® on Hemostasis After Transradial Artery Access
Brief Title: Hemostasis With QuikClot® Radial® Pad Versus TR Band® After Transradial Artery Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Healthcare System (Other)
Collaborators: Z-Medica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QuikClot300
Record Dates: First submitted 2018-05-02; First posted 2018-05-24 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
Keywords: Transradial Access; Hemostasis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomized Controlled prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Arm 1 (No Intervention): TR Band inflated with 10 mL of air, followed by gradual weaning over the subsequent 60 minutes.
- Arm 2 (Experimental): QC pad with a Coban bandage to hold the pad in place to achieve hemostasis.
  Interventions: Device: Quikclot Radial (QC) Pad
- Arm 3 (Experimental): QC pad with a Tegaderm dressing to hold the pad in place to achieve hemostasis.
  Interventions: Device: Quikclot Radial (QC) Pad
- Arm 4 (Experimental): QC pad with a TR Band to hold the pad in place to achieve hemostasis.
  Interventions: Device: Quikclot Radial (QC) Pad

INTERVENTIONS:
Device: Quikclot Radial (QC) Pad — The QC pad will be applied over the radial artery access site covered with either a Coban™ bandage, a Tegaderm™ dressing, or a TR Band after TRA.
  Arms: Arm 2; Arm 3; Arm 4

SUMMARY:
To evaluate the efficacy and safety of the QuikClot® Radial® pad on hemostasis after transradial access (TRA), compared to the standard of care TR Band®, to hopefully develop a safe and efficacious technique to achieve more rapid patent hemostasis after TRA, and improve patient care by optimizing radial hemostasis management.

DETAILED DESCRIPTION:
The QuikClot® Radial® (QC) pad will be applied over the radial artery access site covered with either a Coban™ bandage or a Tegaderm™ dressing after TRA. Firm manual compression will then be applied over the QC pad after the sheath is removed for 5 minutes. The Coban™ cohort will then have the Coban™ bandage removed after an additional 25 minutes, then be covered with a Tegaderm™ dressing. The Tegaderm™ only cohort will be closely observed for 25 minutes after release of manual pressure. Both cohorts will remove the Tegaderm™ dressing the following morning.

Consented subjects will be randomly assigned in the cardiac cath lab upon completion of their procedure into one of the following arms:

Arm 1 - Standard of Care with a TR Band®

Arm 2 - QC pad combined with a Coban™ bandage

Arm 3 - QC pad combined with a Tegaderm™ dressing. This arm was stopped after the enrollment of 73 patients and replaced by the QC/TR Band® arm

Arm 4- QC pad was applied on the radial arterial access site with 30 minutes of compression under a TR Band® inflated with 8-10 mL of air. Then the TR Band® was removed, leaving the QC pad covered with a Tegaderm™ dressing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing cardiac catheterization (CC) and/or percutaneous coronary intervention (PCI) via the radial artery as part of their standard of care treatment
2. Patients able and willing to give written informed consent
3. Patient > 18 years of age

Exclusion Criteria:

1. Patients presenting with acute ST-segment elevation myocardial infarction (STEMI)
2. Oral anticoagulation therapy as described below:

   1. If on a DOAC (direct-acting oral anticoagulants - ie dabigatran, rivaroxaban, apixaban, edoxaban), patients will be excluded if DOAC taken within 48 hours and eGFR > 30 ml/min or DOAC taken within 72 hours and eGFR < 30 ml/min.
   2. If the patient is on warfarin, excluded if INR > 1.5
3. Liver Failure
4. Life-threatening illness that the patient would not be expected to live more than 6 months post-procedure
5. Major unanticipated event in the cardiac cath lab (i.e. cardiac arrest) of an already consented patient, but before randomization, where the operator believes participation in this trial is now inappropriate.
6. Thrombocytopenia, with a platelet count of < 75,000.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Roberts, MD, Principal Investigator — Memorial Healthcare System
Locations (1):
- Memorial Healthcare System, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants ≥ 18 years of age willing to give written informed consent were randomized immediately after the completion of the procedure at the cath lab using the randomization sequence.
Pre-assignment Details: Patients less than 18 years old, acute ST segment elevation myocardial infarction, pregnancy, inability to consent, inability or refusal to allow a follow-up visit or telephone call one business day after the procedure, and arterial access using an ulnar or femoral approach were excluded.
Groups:
- Arm 1: Patients randomly assigned to this arm received 60 min of mechanical compression with a TR Band inflated with 10 mL of air, followed by gradual weaning over the subsequent 60 min. 96 patients who had undergone successful radial access were enrolled in this arm.
- Arm 2: Patients randomly assigned to this arm received the QC pad with 5 minutes of manual pressure followed by 25 minutes of light compression with a Coban™ bandage. 100 patients who had undergone successful radial access were enrolled in this arm.
- Arm 3: Patients randomly assigned to this arm received the QC pad with 5 min of manual pressure followed by a Tegaderm™ dressing. 73 subjects who had undergone successful radial access were enrolled in this arm.
- Arm 4: Patients were assigned to this arm received the QC pad under a TR Band with 30 minutes of compression by the inflated TR Band®. 86 patients who had undergone successful radial access were enrolled in this arm.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 96 | 100 | 73 | 86
Completed | 96 | 100 | 73 | 86
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TR Band: Patients randomly assigned to this arm received 60 min of mechanical compression with a TR Band inflated with 10 mL of air, followed by gradual weaning over the subsequent 60 min. 96 patients who had undergone successful radial access were enrolled in this arm.
- QC/Coban Bandage: Patients randomly assigned to this arm received the QC pad with 5 minutes of manual pressure followed by 25 minutes of light compression with a Coban™ bandage. 100 patients who had undergone successful radial access were enrolled in this arm.
- QC/Trgaderm Dressing: Patients randomly assigned to this arm received the QC pad with 5 min of manual pressure followed by a Tegaderm™ dressing. 73 subjects who had undergone successful radial access were enrolled in this arm.
- QC/TR Band: Patients were assigned to this arm received the QC pad under a TR Band with 30 minutes of compression by the inflated TR Band®. 86 patients who had undergone successful radial access were enrolled in this arm.
- Total: Total of all reporting groups
Arm/Group | TR Band | QC/Coban Bandage | QC/Trgaderm Dressing | QC/TR Band | Total
Number analyzed (Participants) | 96 | 100 | 73 | 86 | 355
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (15.3) | 65.2 (11.4) | 67.1 (13.3) | 64.3 (13.8) | 65.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 19 | 19 | 89
  Male | 70 | 75 | 54 | 67 | 266
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 18 | 17 | 10 | 13 | 58
  Asian | 2 | 4 | 1 | 2 | 9
  Other | 1 | 0 | 0 | 4 | 5
  White | 75 | 79 | 62 | 67 | 283
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (6.5) | 30.3 (7.3) | 29.4 (6.2) | 30.1 (8.5) | 29.9 (7.1)
Hypertension [Count of Participants; unit: Participants] | 80 | 81 | 62 | 69 | 292
Diabetes mellitus [Count of Participants; unit: Participants] | 42 | 40 | 30 | 32 | 144
Dyslipidemia [Count of Participants; unit: Participants] | 62 | 71 | 52 | 59 | 244
Family history of CAD [Count of Participants; unit: Participants] | 1 | 3 | 3 | 6 | 13
Aspirin use [Count of Participants; unit: Participants] | 88 | 90 | 71 | 70 | 319
Oral anticoagulant [Count of Participants; unit: Participants] | 9 | 12 | 11 | 7 | 39

OUTCOME MEASURES:

1. Primary Outcome: Initial Successful Hemostasis
Description: Initial successful hemostasis is defined as no evidence of external bleeding from the TRA puncture site or expanding hematoma of the forearm after completion of the above described TR Band® and QuikClot® Radial® pad protocols, without the need for reinflation of air in the TR Band® or reapplication of manual pressure over the QuikClot® Radial® pad secured with either a Coban™ bandage or Tegaderm™ dressing, or use of manual compression over the arteriotomy site.
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Standard of care TR Band
- Arm 2: QC/Coban bandage
- Arm 3: QC/Tegaderm dressing
- Arm 4: QC/TR Band
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 96 | 100 | 73 | 86
Participants | 85 | 88 | 51 | 74
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Other; p = 0.906, Chi-squared; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.89 to 1.11]
Statistical Analysis 2: Comparison: Arm 1 vs Arm 3; Test type: Other; p = 0.002, Chi-squared; Risk Ratio (RR) = 1.27, 95% CI 2-sided [1.09 to 1.53]
Statistical Analysis 3: Comparison: Arm 1 vs Arm 4; Test type: Other; p = 0.613, Chi-squared; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.86 to 1.09]

2. Primary Outcome: Total Time to Hemostasis
Description: Total time to hemostasis was calculated as the time needed from sheath removal to achieving complete hemostasis. All additional protocol-directed recompression and/or weaning times needed to obtain complete hemostasis were added to calculate the total time to hemostasis.
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 96 | 100 | 73 | 86
minutes | 131.5 (29.8) | 33.3 (9.6) | 10.9 (20.4) | 37.2 (17.3)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -98.5
Statistical Analysis 2: Comparison: Arm 1 vs Arm 3; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -120.6
Statistical Analysis 3: Comparison: Arm 1 vs Arm 4; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -94.3

3. Secondary Outcome: Radial Artery Occlusion (RAO)
Description: RAO will be assessed one hour after completed hemostasis, using the reverse Barbeau's test.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 96 | 100 | 73 | 86
Participants | 5 | 4 | 4 | 3
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Other; p = 0.744, Fisher Exact; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.23 to 2.57]
Statistical Analysis 2: Comparison: Arm 1 vs Arm 3; Test type: Other; p > 0.999, Fisher Exact; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.31 to 3.41]
Statistical Analysis 3: Comparison: Arm 1 vs Arm 4; Test type: Other; p = 0.724, Fisher Exact; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.18 to 2.46]

4. Secondary Outcome: Forearm Hematoma (EASY Classification)
Description: The forearm hematoma development is defined according to the EASY (Early Discharge After Transradial Stenting of Coronary Arteries) classification.
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Standard of care
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 96 | 100 | 73 | 86
Participants | 6 | 9 | 5 | 8
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Other; p = 0.594, Fisher Exact; Risk Ratio (RR) = 1.44, 95% CI 2-sided [0.56 to 3.76]
Statistical Analysis 2: Comparison: Arm 1 vs Arm 3; Test type: Other; p > 0.999, Fisher Exact; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.37 to 3.26]
Statistical Analysis 3: Comparison: Arm 1 vs Arm 4; Test type: Other; p = 0.581, Fisher Exact; Risk Ratio (RR) = 1.45, 95% CI 2-sided [0.55 to 3.88]

5. Secondary Outcome: Incidence of Pain/Numbness of the Forearm
Description: Self-reported pain/numbness was evaluated using a verbal numeric rating scale (VNRS), ranging from 0 for no pain to 10 for the worst pain, one hour after hemostasis was obtained.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 96 | 100 | 73 | 86
Participants | 5 | 10 | 8 | 9
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Other; p = 0.284, Fisher Exact; Risk Ratio (RR) = 1.92, 95% CI 2-sided [0.71 to 5.22]
Statistical Analysis 2: Comparison: Arm 1 vs Arm 3; Test type: Other; p = 0.243, Fisher Exact; Risk Ratio (RR) = 2.10, 95% CI 2-sided [0.75 to 5.9]
Statistical Analysis 3: Comparison: Arm 1 vs Arm 4; Test type: Other; p = 0.266, Fisher Exact; Risk Ratio (RR) = 2.01, 95% CI 2-sided [0.74 to 5.54]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: pseudoaneurysm or any other vascular complications during the observation period. Access site bleeding requires surgery or special medical intervention.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/100 | 0/73 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/100 | 0/73 | 0/86
Other Adverse Events (participants affected / at risk) | 0/96 | 0/100 | 0/73 | 0/86

LIMITATIONS AND CAVEATS:
This is a single-center study that used the QuikClot® Radial® Pad for hemostasis after radial artery access. There is limited past data on the efficacy of this product that has not been widely used in the past for radial artery hemostasis. The points of view expressed in this report are solely those of the investigative team and do not necessarily represent those of their affiliated organizations or the sponsor, and do not provide a concrete basis for the development of practice guidelines.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT03535597/Prot_SAP_000.pdf